CLINICAL TRIAL: NCT05962840
Title: A Prospective, Randomized, Single-blinded Placebo-controlled, Single Center Clinical Study of the Efficacy and Safety for Rituximab Combined With Telitacicept in the Treatment of ANCA-associated Vasculitis
Brief Title: Efficacy and Safety for Rituximab Combined With Telitacicept in the Treatment of ANCA-associated Vasculitis (TTCAAVREM)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSTAR-K2956
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: ANCA Associated Vasculitis
Keywords: Telitacicept; relapse rate; remission maintain treatment
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — telitacicept

STUDY DESIGN:
Intervention Model Description: prospective, randomized, single-blinded, placebo-controlled, pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo arm (Placebo Comparator): Patients with active AAV will be treated with Rituximab and glucocorticoid to induce remission. And the placebo of Telitacicept would be given 80 mg every week subcutaneously for 12 months. Glucocorticoid would be tapered as recommended by 2022 EULAR AAV recommendation (as protocol of PEXIVAS study)
  Interventions: Other: Placebo of Telitacicept
- Telitacicept treatment arm (Experimental): Patients with active AAV will be treated with Rituximab and glucocorticoid to induce remission. And the Telitacicept would be given 80 mg every week subcutaneously for 12 months. Glucocorticoid would be tapered as recommended by 2022 EULAR AAV recommendation (as protocol of PEXIVAS study)
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — Patient will be treated with Telitacicept (Taiai the commercial name) 80 mg every week subcutaneously for 12 months
  Other Names: Taiai for commercial name
  Arms: Telitacicept treatment arm
Other: Placebo of Telitacicept — Patient will be treated with placebo of Telitacicept (Taiai the commercial name) 80 mg every week subcutaneously for 12 months
  Arms: Placebo arm

SUMMARY:
This study is a prospective, open-labelled, randomized, controlled, single-center clinical trial. The aim of this study is to investigate the remission rate of patients treated with Telitacicept combined with Rituximab in remission-induction and Telitacicept alone in remission-maintain treatment.

DETAILED DESCRIPTION:
Background: The basic theme of AAV is relapse and remission. The maintenance therapy of AAV aimed to reduce or prevent relapse is very challenge. Although many medications have been used for the maintenance of AAV, Telitacicept (a BAFF/APRIL dual-target-inhibitor, which has been proved to be effect in treatment of SLE) has not been studied yet. One study tested the efficacy of Belimumab in the maintenance therapy for AAV. When taken Rituximab as remission-induction treatment, no relapse was observed. However, the sample size of this study is small, and the Belimumab, as a BAFF inhibitor, was not been proved to have effect on APRIL.

Many experiences have been accumulated about the efficacy and safety of Telitacicept in Chinese patients with rheumatic diseases. But there is no study to show its effectiveness in the reduction of the relapse of AAV in China. In this study, we take Telitacicept as maintain treatment in AAV patients who receive Rituximab as remission-induction treatment, to verify the effectiveness of Telitacicept in maintenance therapy of AAV.

Objectives: To investigate the effectiveness of Telitacicept in reducing relapse rate by using from remission-induction treatment combined with Rituximab to maintenance treatment of AAV.

Study Design: This is a prospective, randomized, open-label, control, pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 to 65 years, both genders can be included.
2. Patients who are newly diagnosed or relapsing granulomatosis with polyangiitis or microscopic polyangiitis must fulfill the 2022 ACR/EULAR classification criteria of GPA or MPA.
3. Patients have severe active AAV according to the 2021 ACR/vasculitis foundation definition.
4. Patients have to be PR3-ANCA-positive at diagnosis or during the course of their disease.

Exclusion Criteria:

1. Patients who had been treated with Rituximab but had to stop due to adverse events or intolerance.
2. Patients who had other autoimmune diseases.
3. Patients with severe liver dysfunction (defined as the 2-folds elevation of normal upper limit or Child grade III), heart failure or ESRD (eGFR<30ml/min).
4. Patients who are pregnant or have planned for pregnancy in next 2 years.
5. Patients with uncontrolled sever hypertension, diabetes, active bacteria or fungal infection.
6. Patients with active hepatitis virus infection as well as patients who have active mycobacteria infection.
7. Patients with malignancy.
8. Patients who are not eligible according to the judge of the principal investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The time of first relapse during 24 months follow-up of two groups | from inclusion to the end of the study, 24 months in total
  The time from baseline to first relapse(re-appearance of disease with a BVAS >0) of patients during 24 months follow-up of two groups

SECONDARY OUTCOMES:
The time to remission of two groups | from inclusion to the end of the study, 24 months in total
  The time from baseline to remission (disappearance of disease with a BVAS = 0) of patients of two groups
The time from remission to first relapse of two groups | from inclusion to the end of the study, 24 months in total
  The time from remission (disappearance of disease with a BVAS = 0) to first relapse (re-appearance of disease with a BVAS >0) of patients of two groups
The percentage of patients with sustained remission at months 12 and at months 24 of two groups | from inclusion to the end of the study, 24 months in total
  The percentage of patients with sustained remission (disappearance of disease with a BVAS = 0) at months 12 and at months 24 of two groups
The percentage of patients with relapse at months 12 and at months 24 of two groups | from inclusion to the end of the study, 24 months in total
  The percentage of patients with relapse (re-appearance of disease with a BVAS >0), major relapse (re-appearance or worsening of disease with a BVAS >0 and involvement of at least one major organ, a life-threatening manifestation, or both) and minor relapse (re-appearance of disease with a BVAS >0 without involvement of major organ or a life-threatening manifestation) at months 12 and at months 24 of two groups
The rate of adverse events and their severity in both treatment groups during 24 months of the study period. | from inclusion to the end of the study, 24 months in total
  The rate of adverse events and their severity (Severe events were defined as the adverse events of grade 3 or 4, deaths caused by any cause, cancers, side effects that necessitate hospitalization) in both treatment groups during the study period.
The percentage of patients who progress to ESRD at the end of the study | from inclusion to the end of the study, 24 months in total
  The percentage of patients who progress to ESRD at the end of the study
The time of ANCA from positive to negative of two groups | from inclusion to the end of the study, 24 months in total
  The time of ANCA from positive to negative of two groups
The rate of complication of AAV in both treatment groups during 24 months of the study period. | from inclusion to the end of the study, 24 months in total
  The rate of complication of AAV in both treatment groups during 24 months of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, Principal Investigator — Peking Unione Mdecial College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Only patient clincial information coud be released to public